CLINICAL TRIAL: NCT05362942
Title: A Study of Combination of Venetoclax, Hypomethylation Agent and Low-dose Cytarabine as a Salvage Therapy in Patients With Acute Myeloid Leukemia Who Had Relapsed/Refractory Disease or Positive Minimal Residual Disease
Brief Title: Combination of Venetoclax, Hypomethylation Agent and Low-dose Cytarabine as a Salvage Therapy for Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Ning Gao, Principal Investigator, Beijing 302 Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAA-RR&MRD2022V1.0
Record Dates: First submitted 2022-04-20; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Minimal Residual Disease
Keywords: Venetoclax; Hypomethylation agent; Cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — venetoclax; Decitabine; Azacitidine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- venetoclax + Hypomethylation agent + low-dose cytarabine treatment group (Experimental): patients treated with venetoclax combined with decitabine/azacytidine and low-dose cytarabine
  Interventions: Drug: Venetoclax, Decitabine, Azacytidine, Cytarabine

INTERVENTIONS:
Drug: Venetoclax, Decitabine, Azacytidine, Cytarabine — Venetoclax was given at a dose of 400 mg/day for 28 days per cycle. Decitabine was given at a dose of 20 mg/m2/day for 5 days (n=3) or azacytidine (n=8) was given at a dose of 75 mg/m2/day for 7 days at the discretion of the treating physician. Cytarabine was given at a dose of 10 mg/m2 twice daily for 7 days.
  Other Names: Venetoclax (ABT-199, GDC-0199); Decitabine (Dacogen, 5-aza-2-deoxycytidine); Azacitidine (5-Azacytidine, Ladakamycin); Cytarabine (Cytarabine hydrochloride)

SUMMARY:
Although studies are ongoing to evaluate the efficiency and safety of venetoclax-based therapy, alone or in combination with hypomethylation agent or low-dose cytarabine, in relapsed/refractory acute myeloid leukemia, data are scarce and heterogenous. In this study, the investigators aimed to assess safety and response to a new venetoclax-based triple-drug combination regimen (venetoclax + hypomethylation agent + low-dose cytarabine) in acute myeloid leukemia patients who had relapsed/refractory disease or positive minimal residual disease.

DETAILED DESCRIPTION:
Although the promising activity of venetoclax-based therapy is well demonstrated in the treatment of previously untreated elderly or unfit patients with acute myeloid leukemia, there are few data on the efficacy of venetoclax-based salvage therapy in relapsed/refractory patients, which can be difficult to treat. To date, data on venetoclax as monotherapy or in combination with hypomethylation agent or low-dose cytarabine as a salvage regimen in relapsed/refractory AML are scarce and heterogenous. In this study, the investigators aimed to assess safety and efficiency of a new triple-drug combination regimen, venetoclax + hypomethylation agent + low-dose cytarabine, in patients with relapsed/refractory acute myeloid leukemia or persistent positive minimal residual disease in the salvage setting.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years old, voluntarily participate in clinical research and sign an informed consent form and be willing to follow and be able to complete all experimental procedures.
2. The toxic and side effects caused by the last treatment should be recovered.
3. Eastern Cooperative Oncology Group score of 0 to 3 points.
4. The organ function is intact.

   * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤2.5×ULN (Upper Limit of Normal).
   * Creatinine≤1.5×ULN.
   * Bilirubin≤1.5×ULN.
5. Karnofsky≥70.
6. The expected survival period is at least 12 weeks.
7. Non-pregnant, non-breastfeeding women.

Exclusion Criteria:

1. Suffering from other untreated or unrelieved malignant tumors within 2 years.
2. Major surgery, radiotherapy, chemotherapy, biological therapy, immunotherapy, and experimental therapy were performed within 2 weeks of the first medication.
3. Suffering from any other known serious and/or uncontrolled disease (eg, uncontrolled diabetes; cardiovascular disease, including congestive heart failure New York Heart Association [NYHA] Class III or IV, 6 months patients with myocardial infarction and poorly controlled blood pressure); chronic renal failure; or active uncontrolled infection); the investigators considered unsuitable for this clinical trial.
4. Patients who are unwilling or unable to comply with the protocol.
5. Currently being treated with other systemic anti-tumor or anti-tumor research drugs.
6. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | At the end of Cycle 2 (each cycle is 28 days)
  percentage of subjects with complete remission (CR) and incomplete hematologic recovery (CRi)
Complete minimal residual disease (MRD) Response Rate | At the end of Cycle 2 (each cycle is 28 days)
  Percentage of subjects with MRD negative or MRD < 0.01%
MRD Response Rate | At the end of Cycle 2 (each cycle is 28 days)
  Percentage of subjects with MRD < 0.1% detectable by multicolor flow cytometry

SECONDARY OUTCOMES:
Relapse-Free Survival | 24 months
  Time interval from leukemia free state to the first recurrence or death
Overall Survival | 24 months
  Time interval from start of treatment until death or last follow-up
Duration of response | 24 months
  Time interval from morphologic/MRD response to loss of response or death
Adverse events | start of treatment to 2 weeks after end of treatment
  Number of subjects with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-ning Gao, Principal Investigator — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burnett AK. Acute myeloid leukemia: treatment of adults under 60 years. Rev Clin Exp Hematol. 2002 Mar;6(1):26-45; discussion 86-7. doi: 10.1046/j.1468-0734.2002.00058.x. PMID 12060482
- [Background] Breems DA, Van Putten WL, Huijgens PC, Ossenkoppele GJ, Verhoef GE, Verdonck LF, Vellenga E, De Greef GE, Jacky E, Van der Lelie J, Boogaerts MA, Lowenberg B. Prognostic index for adult patients with acute myeloid leukemia in first relapse. J Clin Oncol. 2005 Mar 20;23(9):1969-78. doi: 10.1200/JCO.2005.06.027. Epub 2005 Jan 4. PMID 15632409
- [Background] Burnett A, Wetzler M, Lowenberg B. Therapeutic advances in acute myeloid leukemia. J Clin Oncol. 2011 Feb 10;29(5):487-94. doi: 10.1200/JCO.2010.30.1820. Epub 2011 Jan 10. PMID 21220605
- [Background] Roboz GJ, Rosenblat T, Arellano M, Gobbi M, Altman JK, Montesinos P, O'Connell C, Solomon SR, Pigneux A, Vey N, Hills R, Jacobsen TF, Gianella-Borradori A, Foss O, Vetrhusand S, Giles FJ. International randomized phase III study of elacytarabine versus investigator choice in patients with relapsed/refractory acute myeloid leukemia. J Clin Oncol. 2014 Jun 20;32(18):1919-26. doi: 10.1200/JCO.2013.52.8562. Epub 2014 May 19. PMID 24841975
- [Background] DiNardo CD, Pratz K, Pullarkat V, Jonas BA, Arellano M, Becker PS, Frankfurt O, Konopleva M, Wei AH, Kantarjian HM, Xu T, Hong WJ, Chyla B, Potluri J, Pollyea DA, Letai A. Venetoclax combined with decitabine or azacitidine in treatment-naive, elderly patients with acute myeloid leukemia. Blood. 2019 Jan 3;133(1):7-17. doi: 10.1182/blood-2018-08-868752. Epub 2018 Oct 25. PMID 30361262
- [Background] Wei AH, Strickland SA Jr, Hou JZ, Fiedler W, Lin TL, Walter RB, Enjeti A, Tiong IS, Savona M, Lee S, Chyla B, Popovic R, Salem AH, Agarwal S, Xu T, Fakouhi KM, Humerickhouse R, Hong WJ, Hayslip J, Roboz GJ. Venetoclax Combined With Low-Dose Cytarabine for Previously Untreated Patients With Acute Myeloid Leukemia: Results From a Phase Ib/II Study. J Clin Oncol. 2019 May 20;37(15):1277-1284. doi: 10.1200/JCO.18.01600. Epub 2019 Mar 20. PMID 30892988
- [Background] DiNardo CD, Jonas BA, Pullarkat V, Thirman MJ, Garcia JS, Wei AH, Konopleva M, Dohner H, Letai A, Fenaux P, Koller E, Havelange V, Leber B, Esteve J, Wang J, Pejsa V, Hajek R, Porkka K, Illes A, Lavie D, Lemoli RM, Yamamoto K, Yoon SS, Jang JH, Yeh SP, Turgut M, Hong WJ, Zhou Y, Potluri J, Pratz KW. Azacitidine and Venetoclax in Previously Untreated Acute Myeloid Leukemia. N Engl J Med. 2020 Aug 13;383(7):617-629. doi: 10.1056/NEJMoa2012971. PMID 32786187
- [Background] Bewersdorf JP, Giri S, Wang R, Williams RT, Tallman MS, Zeidan AM, Stahl M. Venetoclax as monotherapy and in combination with hypomethylating agents or low dose cytarabine in relapsed and treatment refractory acute myeloid leukemia: a systematic review and meta-analysis. Haematologica. 2020 Nov 1;105(11):2659-2663. doi: 10.3324/haematol.2019.242826. No abstract available. PMID 33131256
- [Background] Qin T, Youssef EM, Jelinek J, Chen R, Yang AS, Garcia-Manero G, Issa JP. Effect of cytarabine and decitabine in combination in human leukemic cell lines. Clin Cancer Res. 2007 Jul 15;13(14):4225-32. doi: 10.1158/1078-0432.CCR-06-2762. PMID 17634552